CLINICAL TRIAL: NCT03972878
Title: Foodprint 1.0: Metabolic, Hormonal, Inflammatory and Oxidative Post-prandial Responses After Consumption of Confectionary Products
Brief Title: Foodprint 1.0: Physiological Acute Responses After Consumption of Confectionary Products
Acronym: FP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Daniele Del Rio, Professor of Nutrition at Department of Veterinary Science, University of Parma, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FP-1.0
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Glucose, High Blood; Inflammatory Response; Oxidative Stress; Endotoxemia
MeSH Terms: conditions — Endotoxemia

STUDY DESIGN:
Intervention Model Description: The study is a cross-over, randomized intervention trial. Each subject consumed in a randomly order seven foods test with a one-week wash out between different treatments. The portion size of each foods test was calculated in order to provide the same calories.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- control snack (Active Comparator): control snack
  Interventions: Other: control snack
- control cream (Experimental): control spreadable cream
  Interventions: Other: control cream
- cream version 1 (Experimental): control spreadable cream, version 1
  Interventions: Other: cream version 1
- cream version 2 (Experimental): control spreadable cream, version 2
  Interventions: Other: cream version 2
- cream version 3 (Experimental): control spreadable cream, version 3
  Interventions: Other: cream version 3
- control chocolate bar (Experimental): control chocolate bar
  Interventions: Other: control chocolate bar
- chocolate bar version 1 (Experimental): control chocolate bar version 1
  Interventions: Other: chocolate bar version 1

INTERVENTIONS:
Other: control snack — dry fruit snack (200 kcal) + 250 ml water
  Arms: control snack
Other: control cream — commercial spreadable cocoa and hazelnut cream (200 kcal)+ 250 ml water
  Arms: control cream
Other: cream version 1 — commercial spreadable cocoa and hazelnut cream (200 kcal), version 1+ 250 ml water
  Arms: cream version 1
Other: cream version 2 — commercial spreadable cocoa and hazelnut cream (200 kcal), version 2+ 250 ml water
  Arms: cream version 2
Other: cream version 3 — commercial spreadable cocoa and hazelnut cream (200 kcal), version 3+ 250 ml water
  Arms: cream version 3
Other: control chocolate bar — commercial chocolate bar (200 kcal)+ 250 ml water
  Arms: control chocolate bar
Other: chocolate bar version 1 — commercial chocolate bar (200 kcal), version 1+ 250 ml water
  Arms: chocolate bar version 1

SUMMARY:
The composition of a food or a meal consumed plays an important role in the rate of postprandial endocrine and metabolic response, especially if high in fats, sugars and total energy content and a reduction in its entity is related to beneficial effects towards the prevention of several chronical diseases. The physiological postprandial response depends on several factors, both intrinsic, such as natural characteristic of food, and extrinsic, such as the way in which food is processed. This study aims at investigating postprandial hormonal, metabolic, oxidative stress, inflammation and endotoxaemia responses after the consumption of different commercial confectionary products made with different reformulation (ingredients and/or processing techniques).The principal scope of the study is to evaluate the impact of the reformulation of different snacks on postprandial responses. The investigators therefore designed a randomized controlled crossover trial, in which 15 healthy volunteers will consume different isocaloric confectionary products (snacks) and their related reformulation (total products number = 6) and a reference snack. Venous blood samples will be collected until 4-h after meal consumption. In order to evaluate postprandial hormonal, metabolic, oxidative stress, inflammation and endotoxaemia responses several markers will be evaluate:

* metabolic substrates: glucose; Triglycerides and NEFA;
* hormones: insulin; c-peptide; GLP-1, GIP, leptin, ghrelin, PYY;
* markers of inflammation: IL-6, IL-8, IL-10, IL-17, TNF-α, hsCRP, MCP-1;
* markers of oxidative stress and antioxidant capacity: GSH, FRAP;
* endotoxaemia: lipopolysaccharides (LPS).

These results will contribute to a detailed evaluation of the effects of reformulation on physiological events after meal consumption, leading to clarify if these variations in ingredients and/or processing techniques can modify postprandial responses, making them more similar to those originated from the reference snack.

DETAILED DESCRIPTION:
Meal consumption, especially if high in fats, sugars and total energy content, leads to a transient rise in blood glucose and lipids. The extent of glycemic and lipidemic postprandial responses have been linked to the progression of cardiovascular and other chronic degenerative diseases, such as type 2 diabetes and Alzheimer through a substantial increase in oxidative stress, systemic inflammation, and endothelial dysfunction. In addition, some studies have shown that consuming a high fat meal is associated with a postprandial increase in plasma and serum endotoxin concentrations in humans. LPS, lipopolysaccharide, is considered a major predisposing factor for inflammation-associated diseases such as atherosclerosis, sepsis and obesity. Therefore, following a correct dietary model may be beneficial in order to limit postprandial excursion and to modulate hormonal responses involved in satiety.

The physiological postprandial response depends on several factors, both intrinsic, such as natural characteristic of food, and extrinsic, such as the way in which food is processed. Thus, the present study aims at evaluating if the reformulation of some commercial confectionery products can lead to an improvement of the nutritional profile, through a decrease of postprandial metabolic and hormonal, oxidative stress, inflammation and endotoxaemia responses in comparison with commercial confectionery products (snacks).

ELIGIBILITY:
Inclusion Criteria:

- Healthy male and female adult subjects

Exclusion Criteria:

* BMI > 30 kg/m2
* Metabolic disorders (diabetes, hypertension, dyslipidemia, glucidic intolerance)
* Chronic drug therapies for any pathologies (including psychiatric diseases)
* Dietary supplements affecting metabolism of glucose and lipid
* Celiac disease
* Pregnancy or lactation
* Lactose intolerance
* Food allergies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
IAUC postprandial blood glucose | 0 (fasting), 15, 30, 45, 60, 90, 120, 180, 240 minutes
  Incremental area under the curve of blood glucose postprandial response (IAUC)

SECONDARY OUTCOMES:
Postprandial response for blood glucose | 0 (fasting), 15, 30, 45, 60, 90, 120, 180, 240 minutes
  incremental blood glucose concentration at each timepoint of the curve
IAUC postprandial blood hormones (insulin, c-peptide, ghrelin, Glucagon-like peptide 1 (GLP-1), Gastric inhibitory peptide (GIP), peptide YY (PYY), leptin) | 0 (fasting), 15, 30, 45, 60, 90, 120, 180, 240 minutes
  Incremental area under the curve for blood insulin postprandial response (IAUC)
Postprandial response for blood hormones (insulin, c-peptide, ghrelin, Glucagon-like peptide 1 (GLP-1), Gastric inhibitory peptide (GIP), peptide YY (PYY), leptin) | 0 (fasting), 15, 30, 45, 60, 90, 120, 180, 240 minutes
  incremental blood insulin concentration at each timepoint of the curve
IAUC postprandial blood lipids triglycerides (TAG) and non esterified fatty acid (NEFA) | 0 (fasting), 30, 60, 90, 120, 180, 240 minutes
  Incremental area under the curve for blood TAG and NEFA postprandial response (IAUC)
Postprandial response for blood lipids triglycerides (TAG) and non esterified fatty acid (NEFA) | 0 (fasting), 30, 60, 90, 120, 180, 240 minutes
  incremental blood TAG and NEFA concentration at each timepoint of the curve
IAUC postprandial blood inflammatory markers (IL-6, IL-8, IL-10, IL-17, TNF-α, hsCRP, MCP-1) | 0 (fasting), 60, 90, 120, 180, 240 minutes
  Incremental area under the curve for blood inflammatory markers (IL-6, IL-8, IL-10, IL-17, TNF-α, hsCRP, MCP-1) postprandial response (IAUC)
Postprandial response for blood inflammatory markers (IL-6, IL-8, IL-10, IL-17, TNF-α, hsCRP, MCP-1) | 0 (fasting), 60, 90, 120, 180, 240 minutes
  incremental blood inflammatory markers (IL-6, IL-8, IL-10, IL-17, TNF-α, hsCRP, MCP-1) concentration at each timepoint of the curve
IAUC postprandial blood oxidative stress related markers glutathione (GSH) and antioxidant capacity (Ferric ion reducing antioxidant power (FRAP)) | 0 (fasting), 60, 90, 120, 180, 240 minutes
  Incremental area under the curve for blood oxidative stress related markers glutathione (GSH) and antioxidant capacity (Ferric ion reducing antioxidant power (FRAP))
Postprandial response for blood oxidative stress related markers glutathione (GSH) and antioxidant capacity (Ferric ion reducing antioxidant power (FRAP)) | 0 (fasting), 60, 90, 120, 180, 240 minutes
  incremental blood oxidative stress related markers glutathione (GSH) and antioxidant capacity (Ferric ion reducing antioxidant power (FRAP)) concentration at each timepoint of the curve
IAUC postprandial blood endotoxemia (Lipopolysaccharides (LPS)) | 0 (fasting), 60, 90, 120, 180, 240 minutes
  Incremental area under the curve for LPS
Postprandial response for blood LPS | 0 (fasting), 60, 90, 120, 180, 240 minutes
  incremental blood LPS concentration at each timepoint of the curve

OTHER OUTCOMES:
Postprandial satiety using a 100mm visual analog scale | 0 (fasting), 15, 30, 60, 120, 240 minutes
  Differences in subject-rated satiety using a 100mm visual analog scale (centimeter) Range 0-10 centimeter. Higher are the values of satiety in each timepoints better is the product.
Palatability | 12 minutes (after consumption)
  Palatability using a 100mm visual analog scale (centimeter). Range 0-10 centimeter. Higher is the value of palatability better is the product.
Postprandial gastrointestinal symptoms using a 100mm visual analog scale | 0 (fasting), 15, 30, 60, 120, 240 minutes
  gastrointestinal symptoms using a 100mm visual analog scale (centimeter). range 0-10 centimeter. Lower are the values of gastrointestinal symptoms better is the product.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Parma, Italy

REFERENCES:
- [Background] Emerson SR, Kurti SP, Harms CA, Haub MD, Melgarejo T, Logan C, Rosenkranz SK. Magnitude and Timing of the Postprandial Inflammatory Response to a High-Fat Meal in Healthy Adults: A Systematic Review. Adv Nutr. 2017 Mar 15;8(2):213-225. doi: 10.3945/an.116.014431. Print 2017 Mar. PMID 28298267
- [Background] Erridge C, Attina T, Spickett CM, Webb DJ. A high-fat meal induces low-grade endotoxemia: evidence of a novel mechanism of postprandial inflammation. Am J Clin Nutr. 2007 Nov;86(5):1286-92. doi: 10.1093/ajcn/86.5.1286. PMID 17991637
- [Background] Herieka M, Erridge C. High-fat meal induced postprandial inflammation. Mol Nutr Food Res. 2014 Jan;58(1):136-46. doi: 10.1002/mnfr.201300104. Epub 2013 Jul 12. PMID 23847095
- [Background] O'Keefe JH, Bell DS. Postprandial hyperglycemia/hyperlipidemia (postprandial dysmetabolism) is a cardiovascular risk factor. Am J Cardiol. 2007 Sep 1;100(5):899-904. doi: 10.1016/j.amjcard.2007.03.107. Epub 2007 Jun 26. PMID 17719342
- [Background] Treib J, Haass A, Kiessig ST, Woessner R, Grauer MT, Schimrigk K. Tick-borne encephalitis diagnosis in patients with inflammatory changes in the cerebrospinal fluid in a region with very low prevalence. Infection. 1996 Sep-Oct;24(5):400-2. doi: 10.1007/BF01716095. PMID 8923057